CLINICAL TRIAL: NCT02162095
Title: Is Chronic Obstructive Pulmonary Disease a Risk Factor for Cardiovascular Disease?
Brief Title: Is COPD a Risk Factor for Cardiovascular Disease?
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: SNCTP000000995
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Coronary artery disease; Coronary calcium score
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic obstructive pulmonary disease: Approximately 100 participants with documented chronic obstructive pulmonary disease (post-bronchodilator Forced expiratory volume in 1 second (FEV1)/Forced vital capacity (FVC) < 0.7).
- Control: Approximately 100 participants with exclusion of chronic obstructive pulmonary disease (post-bronchodilator Forced expiratory volume in 1 second (FEV1)/Forced vital capacity (FVC) > 0.7).

SUMMARY:
Patients with chronic obstructive pulmonary disease suffer from significant cardiovascular morbidity and mortality. This study wants to determine whether chronic obstructive pulmonary disease might be a risk factor for coronary atherosclerosis and other cardiac markers independent of conventional cardiovascular risk factors. The study is designed as a retrospective matched case-control study with follow-up via telephone interview.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) suffer from significant cardiovascular morbidity and mortality. Coronary artery disease has often been linked causally to COPD, but the exact pathophysiological mechanisms underpinning this association remain speculative. A retrospective case-control study matching COPD patients and controls one to one for smoking history and conventional cardiovascular risk factors will be performed to study the association between COPD and cardiovascular outcomes. Filling in this knowledge gap may contribute to the understanding of the interplay between COPD and cardiovascular disease.

The objective of this retrospective case-control study is to determine whether COPD might be a risk factor for coronary atherosclerosis, impaired left ventricular ejection fraction, and major adverse cardiovascular events independent of conventional cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* SPECT-CT imaging due to preoperative assessment between 01.01.2007 and 31.07.2013.
* Coronary artery calcium score and left ventricular ejection fraction data available.
* History of smoking (smoker or ex-smoker).
* COPD group: Documented chronic obstructive pulmonary disease (post-bronchodilator FEV1/FVC < 0.7).
* Control group: Exclusion of chronic obstructive pulmonary disease (post-bronchodilator FEV1/FVC > 0.7).

Exclusion Criteria:

* Known coronary artery disease or coronary symptoms (angina pectoris) at the time of the SPECT-CT investigation.
* Known congenital or structural heart disease.
* Previous heart transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a history of smoking underdoing SPECT-CT imaging due to preoperative assessmentat the University Hospital Zurich between 01.01.2007 and 31.07.2013.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Coronary calcium score in cardiac computed tomography | Up to one month
  Retrospective assessment of SPECT-CT imaging data at the University Hospital Zurich.

SECONDARY OUTCOMES:
Left ventricular ejection fraction in single-photon emission computed tomography | Up to one month
  Retrospective assessment of SPECT-CT imaging data at the University Hospital Zurich.
Major adverse cardiovascular events | Up to three months
  Follow-up via telephone interview for major adverse cardiovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Canton of Zurich, Switzerland